CLINICAL TRIAL: NCT05157880
Title: Recovering Together: Building Resiliency in Dyads of Patients With an Acute Brain Injury Admitted to the Neuroscience Intensive Care Unit and Their Informal Caregivers
Brief Title: Building Resiliency in Dyads of Patients With an ANI Admitted to the Neuro-ICU and Their Informal Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Associate Professor/Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021P001943
Record Dates: First submitted 2021-10-28; First posted 2021-12-15 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-06

CONDITIONS: Acute Neurological Injury; Emotional Distress
Keywords: Neurological Injury; Emotional Distress; Dyadic Intervention
MeSH Terms: conditions — Trauma, Nervous System

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Patient-Caregiver Dyads (Experimental): There will be 6 sessions with 2 general sessions delivered in person at bedside in the NICU (or virtual depending on COVID and discharge status) and 4 tailored specific sessions (chosen from by the dyads from 6 available modules) to be delivered via live video using Zoom. Content will be primarily skills.
  Interventions: Behavioral: Recovering Together
- Control Patient-Caregiver Dyads (Active Comparator): There will be 6 sessions with 2 general sessions delivered in person at bedside in the NICU (or virtual depending on COVID and discharge status) and 4 tailored specific sessions (chosen from by the dyads from 6 available modules) to be delivered via live video using Zoom. Content will be primarily educational.
  Interventions: Behavioral: Recovering Together

INTERVENTIONS:
Behavioral: Recovering Together — In the skills-based intervention group, sessions focus on developing skills to cope and manage ANI related stressors. The intervention will be tailored consistent with AHA recommendations for ANI skills-based interventions and will include 2 general and 4 specific modules. It is anticipated that the intervention will have 6 sessions with 2 general sessions delivered, in person if possible, within the NICU, or through live video using Zoom if patients leave the hospital before sessions occur, and 4 tailored specific sessions (chosen from by the dyads from 6 available modules) to be delivered via live video using Zoom.
  Other Names: Skills-based intervention
  Arms: Experimental Patient-Caregiver Dyads
Behavioral: Recovering Together — Those in the educational program will receive general health information that mimics the skills-based intervention, but without teaching any of the resiliency or interpersonal communication skills that are hypothesized to be responsible for improvement in emotional distress. There will also be 6 sessions, 2 in-person dyadic visits in the NICU and 4 dyadic virtual visits following discharge. The educational program group will not have the opportunity to specify which modules they would like to take; the modules will be predetermined. All participants will receive medical care as determined by their medical team.
  Other Names: Educational program
  Arms: Control Patient-Caregiver Dyads

SUMMARY:
The purpose of the present investigation is to test the efficacy of a brief (6 sessions) dyadic (patient and caregiver together) intervention to prevent chronic emotional distress in at risk dyads admitted to a Neuroscience Intensive Care Unit with an acute brain injury. Through this study, we seek to solve the unmet need of preventing chronic emotional distress in Neuroscience Intensive Care Unit (NICU) dyads through a feasible, acceptable and credible program, and ideally improve the recovery trajectory and dyads' overall quality of life.

DETAILED DESCRIPTION:
The goals of this study are to: 1) demonstrate the efficacy of Recovering Together for improving self-reported emotional distress (primary outcome), and post traumatic stress, mindfulness, coping, social support and other relevant outcomes (secondary outcomes); and 2) assess mechanisms (mediators and moderators) of improvement after intervention. We will enroll and randomly assign 194 at risk dyads (97 per study group) to receive either the active intervention or educational control. The trial is single blinded (assessors, patients and staff). The trial will take place at the Massachusetts General Hospital NICU using our established methodology successfully implemented during the R21 pilot study. Study clinicians will deliver 6, 30 minute sessions of active intervention or educational control (2 at bedside and 4 via live video after discharge) to each patient-caregiver dyad. All participants will complete measures at baseline, after completion of program (6 weeks) and 3 months later. They will also complete measures of emotional distress weekly, as well as measures assessing home practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English fluency and literacy
* Patient with an informal caregiver available and willing to participate
* Hospitalized with any ANI within 6 weeks (patient) OR informal caregiver of a patient currently admitted with any ANI
* Patient and/or caregiver exhibit emotional distress on screening (using HADS D and/or HADS A scores > 7)

Exclusion Criteria:

* Permanent cognitive impairment (including severe hearing impairment) or aphasia that makes participation impossible
* Short form of Mini-Mental State Exam (SMMSE) score <4 (If SMMSE <4, nursing team decides whether or not the patient can meaningfully participate)
* Glasgow Coma Scale (GCS) score <10
* Terminal diagnosis
* Lack of access to internet and/or a device with a camera
* Current untreated or unstable severe mental health conditions like bipolar disorder, schizophrenia, or active substance use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional Distress | 0 weeks, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 3 months
  Hospital Depression and Anxiety Scale total score (HADS); 0-21 for each subscale (anxiety and depression), higher scores indicate greater anxiety or depression

SECONDARY OUTCOMES:
Change in Post-Traumatic Stress | 0 weeks, 6 weeks, 3 months
  Post-Traumatic Stress Disorder Checklist - Specific Event (PCL-S); 17-85, higher scores indicate greater post-traumatic stress
Change in Resiliency Factors (Mindfulness - curiosity and de-centering) | 0 weeks, 6 weeks, 3 months
  Toronto Mindfulness Scale-Trait (TMS-Trait); 0-52, higher scores indicate greater perceived mindfulness (specifically curiosity and de-centering)
Change in Resiliency Factors (Mindfulness) | 0 weeks, 6 weeks, 3 months
  Cognitive and Affective Mindfulness Scale (CAMS); 12-48, higher scores indicate greater perceived mindfulness
Change in Resiliency Factors (Individual Coping) | 0 weeks, 6 weeks, 3 months
  Measure of Current Status Part A (MOCS-A); 0-52; higher scores indicate greater perceived ability to cope
Change in Resiliency Factors (Dyadic Coping) | 0 weeks, 6 weeks, 3 months
  Dyadic Coping Inventory (DCI); 35-175; higher scores indicate greater perceived coping in the context of a relationship
Change in Interpersonal Factors (perceived social support) | 0 weeks, 6 weeks, 3 months
  Interpersonal Support Evaluation List-12 (ISEL-12); 0-48, higher scores indicate greater perceived social support
Change in Interpersonal Factors (avoidant or anxious communication) | 0 weeks, 6 weeks, 3 months
  Experiences in Close Relationships Scale short form (ECR-S); 7-42, higher scores indicate greater avoidant or anxious communication
Change in Interpersonal Factors (dyadic strain and positive interpersonal interactions) | 0 weeks, 6 weeks, 3 months
  Dyadic Relationship Scale (DRS); Patient version: 10-40, caregiver version: 11-44, dyadic strain subscale: higher scores indicate greater levels of strain, positive dyadic interaction subscale: higher scores indicate greater levels of positive interaction

OTHER OUTCOMES:
Demographic Factors (potential moderators) | 0 weeks
  Age; biological sex; gender; race/ethnicity; educational level; employment status; occupation; income; marital status; prior ANI status; mental health history; psychotropic medications; medical comorbidities; satisfaction with medical staff (analog scale 0-10)
Change in Independence in activities of daily living (potential moderator) | 0 weeks, 6 weeks, 3 months
  Barthel Score; 0-100, higher scores indicate greater independence
Change in Degree of disability or dependence (potential moderator) | 0 weeks, 6 weeks, 3 months
  Modified Rankin; 0-6, higher scores indicate greater disability

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital (MGH), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vranceanu AM, Woodworth EC, Kanaya MR, Bannon S, Mace RA, Manglani H, Duarte BA, Rush CL, Choukas NR, Briskin EA, Cohen J, Parker R, Macklin E, Lester E, Traeger L, Rosand J; Neuro-ICU Recovering Together Team; Grunberg VA. The Recovering Together study protocol: A single-blind RCT to prevent chronic emotional distress in patient-cargiver dyads in the Neuro-ICU. Contemp Clin Trials. 2022 Dec;123:106998. doi: 10.1016/j.cct.2022.106998. Epub 2022 Nov 8. PMID 36368480